CLINICAL TRIAL: NCT04414904
Title: Determining the Reproductive Health of Men Post-COVID-19 Infection
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain approval
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH5998
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Infertility, Male; Testosterone Deficiency
Keywords: infertility; hypogonadism
MeSH Terms: conditions — Infertility, Male; Infertility; Hypogonadism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm DNA fragmentation testing only. No sequencing of human genomic DNA will take place.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: * Men 18-50 years of age
  * Already attending hospital for another reason
  * High risk of prior COVID-19 infection:
    * EITHER Prior positive COVID-19 PCR test result
    * OR history suggestive of COVID-19 illness
  Interventions: Other: Exposure: Covid-19 infection
- Control Group: * Men 18-50 years of age
  * Already attending hospital for another reason
  * Low risk of prior COVID-19 infection:
    * EITHER Negative positive COVID-19 PCR test result within last 4 weeks
    * OR no history suggestive of COVID-19 illness

INTERVENTIONS:
Other: Exposure: Covid-19 infection — Previous history of COVID-19 infection.
  Groups: Case group

SUMMARY:
Study rationale

1. An increasing proportion of the worldwide population is being infected with COVID-19.
2. There are ongoing and currently unanswered safety concerns about the effects of COVID-19 on reproductive health.
3. It will be immensely reassuring to rapidly report that COVID-19 has no detectable effects on male endocrine or sperm function. Conversely, if COVID-19 does impair male reproductive health, appropriate screening can be performed in couples trying to conceive, and further research can be undertaken.
4. The proposed study will be simple, rapid, and authoritative for the UK and worldwide.

DETAILED DESCRIPTION:
Male infertility results from impaired sperm function, and account for half of all infertility. Fertility services have been reported to cost £325M annually in the UK(4) (REF). Testosterone deficiency is one of the most common hormonal problems affecting men, leading to osteoporosis, type 2 diabetes, obesity and depression(5).

Concerns have been raised about the potential effects of COVID-19 on male reproductive dysfunction (male infertility and testosterone deficiency). A recent study has suggested that COVID-19 may enter human cells by binding to receptors (special gates on cells that recognise a specific molecule) for angiotensin converting enzyme 2 (ACE2)(6) . ACE2 receptors are found at very high levels in the testes. Within the testes, ACE2 is found on developing sperm, the 'nurse cells' that help the sperm grow (Sertoli cells), and also on Leydig cells which are needed to make the male sex hormone testosterone. In summary, this evidence suggests that there is a plausible link why COVID-19 would cause male infertility and testosterone deficiency.

All fertility treatment in the UK is regulated by the Human Fertility and Embryology Authority (HFEA). The HFEA has prohibited on all non-cancer fertility treatment in the UK between April 15th and May 12th 2020 due to the COVID-19 epidemic. It is important to rapidly screen and report whether COVID-19 has any obvious effects in causing male infertility and testosterone deficiency. It must be noted that a recent study(1) reported that COVID-19 is not spread by human semen and therefore, semen processing should not risk staff to COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Men 18-50 years of age
* Already attending hospital for another reason
* Low risk of prior COVID-19 infection(EITHER Negative positive COVID-19 PCR test result within last 4 weeks OR no history suggestive of COVID-19 illness)
* High risk of prior COVID-19 infection(EITHER Prior positive COVID-19 PCR test result OR history suggestive of COVID-19 illness)

Exclusion Criteria:

* Men with current symptoms of COVID-19 infection
* Men currently self-isolating as per UK government advice for COVID-19 infection
* Needle-phobia
* Impaired ability to provide full consent to take part in the study
* History of co-morbidity likely to affect male reproductive function e.g. undescended testes, removal of testes, testicular cancer, drugs such as corticosteroids or testosterone therapy.

Ages: 18 Years to 50 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — Male
Study Population: We will be recruiting participants by the following means:
  1. Posters within Imperial College NHS Healthcare trust
  2. Advertisements within newspapers
  3. Online advertisements including in social media websites
  4. Databases held by Imperial College NHS Healthcare trust whereby men have expressed an interest to participate in future research
  5. Patients attending the Andrology Department and other reproductive outpatient clinics at Imperial College NHS healthcare trust
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Semen parameters | 3 visits (up to 75 days apart)
  Sperm concentration (x10^6/ml) between case and control group.
Sperm Parameters | 3 visits (up to 75 days apart)
  Sperm Motility (%) between case and control group.
Sperm Parameters | 3 visits (up to 75 days apart)
  Sperm normal morphology (%) between case and control group.
Hormones measurement | 3 visits (up to 75 days apart)
  Testosterone (nmol/L) between case and control group.
Hormones measurement | 3 visits (up to 75 days apart)
  Follicle Stimulating Hormone(IU/L) between case and control group.
Hormones measurement | 3 visits (up to 75 days apart)
  Luteinising hormone(IU/L) between case and control group.

SECONDARY OUTCOMES:
Seminal Reactive oxygen species | 3 visits (up to 75 days apart)
  Compare seminal reactive oxidative species (RLU/second/10^6sperm) between case and control group.
Sperm DNA fragmentation rate | 3 visits (up to 75 days apart)
  Compare Sperm DNA fragmentation rate (%) between case and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Channa Jayasena, London, Outside U.S./Canada, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Xu X. scRNA-seq Profiling of Human Testes Reveals the Presence of the ACE2 Receptor, A Target for SARS-CoV-2 Infection in Spermatogonia, Leydig and Sertoli Cells. Cells. 2020 Apr 9;9(4):920. doi: 10.3390/cells9040920. PMID 32283711
- [Background] Wang S, Zhou X, Zhang T, Wang Z. The need for urogenital tract monitoring in COVID-19. Nat Rev Urol. 2020 Jun;17(6):314-315. doi: 10.1038/s41585-020-0319-7. PMID 32313110
- [Background] Hackett G, Kirby M, Edwards D, Jones TH, Rees J, Muneer A. UK policy statements on testosterone deficiency. Int J Clin Pract. 2017 Mar;71(3-4):e12901. doi: 10.1111/ijcp.12901. Epub 2017 Mar 20. PMID 28318076
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- See also: The state of the fertility sector 2017-2018 — http://www.hfea.gov.uk
- See also: Reference 1 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7164916/